CLINICAL TRIAL: NCT02512536
Title: Do Ultrasound Guided Botulinum A Injections Relieve Pain in Rotator Cuff Arthropathy?
Brief Title: Does Botulinum A Toxin Help With Pain From Rotator Cuff Arthropathy?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510150
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Intervention:
  Subjects receiving a single ultrasound scan guided injection of Botulinum Toxin type A into the supraspinatus muscle belly.
  Drug: Dysport 300 units im. One single injection over course of study.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Ultrasound scan guided injection into supraspinatus muscle belly with Botulinum Toxin Type A
  Other Names: Dysport

SUMMARY:
Rotator cuff arthropathy is a cause of shoulder arthritis which is a common condition seen both in primary and secondary care. It is a painful condition, with significant disability. Specialist shoulder replacements have found acceptance within the trust, nationally and internationally although there are high complication rates. There is however a significant cost difference (fifty fold) between a reverse total shoulder replacement and a botox injection, and to date there have been no randomised control trials, or any registered, comparing the use of a botox injection for pain relief in cuff arthropathy versus no treatment. If there is a significant clinical difference in the pain outcomes between the two, this could result in significant savings to the NHS and the taxpayer as a whole. If high levels of pain relief could be predictably obtained using Botulinum A toxin injections then potentially patients could avoid the need for surgery.

DETAILED DESCRIPTION:
Null Hypothesis This is a pilot / feasability study. The null hypothesis is that there is no effect on the pain or oxford shoulder scores reported by patients receiving a targeted botulinum A toxin injection in the presence of cuff arthropathy at 6 weeks, 3 months or 6 months compared with the baseline values.

Objectives The aim of this feasability study is to provide the necessary information for the planning of a future trial. It will test the feasibility of running such a trial and provide estimates of the differences in outcome measures and information on resource data.

All potential participants for this study will be identified by an Orthopaedic Shoulder Consultant in the shoulder clinics run at the Royal Devon and Exeter NHS Trust. The patients will be screened for eligibility by a research associate (SG). The eligibility criteria will be that the patient is medically fit for an operation, and has painful rotator cuff arthropathy, that is deemed suitable for intervention by the consultant surgeon. The patients will be informed verbally and in writing about the trial by the research associate and informed consent will be taken.

The participating patients will be allocated to an USS guided botox injection. All patients will be asked to complete a number of questionnaires prior to the injection: the Oxford Shoulder Score (OSS), a Visual Analogue Score (VAS) and the EQ-5D. The range of movement of the shoulder joint will be documented in the usual fashion.

The injections will all be done by Dr Anaspure (Consultant Radiologist) under USS guidance in a standard manner.

After the injection, patients will be reviewed using the range of movement, OSS, a patient satisfaction score and EQ-5D at 6 weeks, 3 months and 6 months post injection. A record will be kept of any complications associated with the treatment. This data will be collected by the research associate, who is independent of either intervention.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria The only eligibility criterion for participation in this study is that the patient is medically fit for an operation and diagnosed with symptomatic rotator cuff arthropathy. They must be able to give informed consent and have evidence of cuff arthropathy on plain radiographs of the affected shoulder.

Exclusion Criteria:

* Exclusion criteria Contra-indications to surgery (defined as severe cardiac impairment, e.g. heart or valve replacement, arrhythmia, previous myocardial infarction; severe respiratory impairment, e.g. chronic obstructive pulmonary disease, asthma that has required hospital admission; any other systemic medical condition that would produce a specific contraindication to a general anaesthetic).

Evidence that the patient would be unable to adhere to trial procedures or complete questionnaires, such as dementia or intravenous drug abuse Note: If a recruited patient requires a contra-lateral shoulder botox injection during the trial period, this second shoulder cannot be included in the study since the result of this intervention would not be independent from the first intervention.

Other exclusion criteria include:

Previous fractures or dislocations of the shoulder. Previous surgery on the affected shoulder. Any neurological or medical condition resulting in spasticity

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Post injection Oxford Shoulder Scores | At 6 weeks, 3 months and 6 months after injection.
  PROM

SECONDARY OUTCOMES:
Pain score | At 6 weeks, 3 months and 6 months after injection.
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Chris Smith, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon and Exeter hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No